CLINICAL TRIAL: NCT03412526
Title: A Phase 2, Single-Center, Open Label Study of Autologous, Adoptive Cell Therapy Following a Reduced Intensity, Non-myeloablative, Lymphodepleting Induction Regimen in Metastatic Ovarian
Brief Title: Adoptive Cell Therapy Following a Reduced Intensity, Non-myeloablative, Lymphodepleting Induction Regimen in Metastatic Ovarian
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Jacob Schachter MD,, Head of Ella Lemelbaum Institute for Immuno- Oncology, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-16-3568-JS-TIL Ovarian
Record Dates: First submitted 2018-01-21; First posted 2018-01-26 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Metastatic Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — fludarabine; Radiation; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACT TIL (Experimental): 1. Reduced Intensity, non-myeloablative, lymphodepleting induction regimen using Fludarabine (25 mg/m2 for 3 days) followed by Total Body Radiation (TBR) (2 Gray as a single treatment) for 1 day
  2. Preparation and administration of unselected or 4-1BB enriched TIL
  3. Bolus high-dose (720,000 IU/kg) IL-2 will be administered to each patient every 8 hours, to tolerance. A maximum of 10 doses will be administered per patient.
  Interventions: Drug: Fludarabine; Radiation: Radiation; Biological: TIL administration; Drug: IL-2

INTERVENTIONS:
Drug: Fludarabine — Reduced intensity, myeloablative, lymphodepleting regimen (25 mg/m2 for 3 days)
Radiation: Radiation — Total Body Radiation (TBR) (2 Gray in a single treatment) for 1 day
Biological: TIL administration — TIL Administration
Drug: IL-2 — bolus high-dose (720,000 IU/kg) IL-2 is administered to the patients every 8 hours, to tolerance. A maximum of 10 doses are given to the patients.

SUMMARY:
Adoptive cell therapy (ACT) with tumor-infiltrating lymphocytes (TILs) in combination with lymphodepletion and high-dose interleukin 2.

Most TIL ACT trials have been conducted as salvage therapy for patients who already had failed numerous treatments; many study participants presented with multiple metastases, frequently in visceral organs and even in the brain. The effectiveness of TIL ACT in eradicating metastatic tumors of the responding patients underlines the value of this immunotherapeutic approach.

Recent developments in the identification and selection of tumor-specific T-cell populations have facilitated the implementation of TIL ACT also in nonmelanoma malignancies. Building on the experience of Ella Lemelbaum Institute, Sheba Medical Center with ACT TIL in the treatment of metastatic melanoma, the Dept. of Oncology, Tel HaShomer has expanded the use of TIL ACT following a reduced intensity, non-myeloablative, lymphodepleting induction regimen to metastatic Melanoma, Ovarian (OC) and Cervical cancer patients. The rationale supporting these studies is to further develop the ACT TIL procedure and expand its applicability to metastatic OC and cervical cancers.

DETAILED DESCRIPTION:
The Sponsor is developing the ex-vivo expanded autologous Tumor Infiltrating Lymphocytes (TIL) as the Investigational Product (IP). Yet, the administration of the TIL cellular product can only be accomplished in the context of an Autologous, Adoptive Cell Therapy (ACT) procedure which is composed of the following steps:

1. Reduced Intensity, non-myeloablative, lymphodepleting induction regimen using Fludarabine (25 mg/m2 for 3 days) followed by Total Body Radiation (TBR) (2 Gray as a single treatment) for 1 day
2. Preparation and administration of unselected or 4-1BB enriched TIL
3. Bolus high-dose (720,000 IU/kg) IL-2 will be administered to each patient every 8 hours, to tolerance. A maximum of 10 doses will be administered per patient.
4. Early-stage follow-up until 30 days post-discharge
5. Late-stage follow-up, such as CT scans, will be carried out four and twelve weeks after TIL administration, and then every 3 months thereafter for the first year after TIL therapy; for the second year and onwards, as clinically indicated.

ELIGIBILITY:
INCLUSION CRITERIA

1. Able to understand and sign the Informed Consent Form.
2. Pathology confirmed epithelial Ovarian/Fallopian Tube/Primary Peritoneal carcinomatosis.
3. For ovarian/peritoneal carcinoma: Platinum- resistant or platinum refractory disease (platinum-resistant disease is defined as disease-progression within 6 months of completion of prior platinum containing regimen, whereas platinum refractory disease is defined as disease progression while on platinum containing regimen or within 3 months from first line, adjuvant chemotherapy).
4. Received and exhausted standard of care therapies for recurrent ovarian cancer and further chemotherapy lines have no proven added value. (For platinum resistant disease, received no more than 3 prior chemotherapy lines, whereas for platinum refractory disease received no more than 2 previous chemotherapy lines).
5. Patients must have at least one lesion that is resectable for TIL generation.
6. Have measurable disease per RECIST 1.1.
7. Patients with one or more brain metastases less than 1 cm each, and any patients with 1 or 2 brain metastases greater than 1 cm must have been treated and stable for 6 weeks.
8. Greater than or equal to 18 years of age.
9. For Patients with child bearing potential, willing to practice birth control from the start of chemotherapy until 120 days after release from the hospital.
10. Life expectancy of greater than three months
11. Performance status of ECOG 0 or 1
12. Adequate organ function defined by lab test results:

    Hematology:

    Absolute neutrophil count greater than 1000/mm3 without support of filgrastim Normal WBC greater than 3000/mm3. Hemoglobin greater than 9.0 g/dL Platelet count greater than 100,000/mm3

    Serology:

    Seronegative for HIV antibody. Seronegative for Hepatitis B or Hepatitis C (patients who recovered from previous infection and have no detected HBSAg or HCV RNA are allowed).

    Chemistry:

    Serum ALT/AST less than three times the upper limit of normal (ULN). Serum creatinine less than or equal to 1.6 mg/dL Total bilirubin no more than 1.5 times the ULN, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3 mg/dL.
13. Negative pregnancy test in women of child bearing potential.
14. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients' toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo). Patients may have undergone minor surgical procedures with the past 3 weeks, as long as all toxicities have recovered to grade 1 or less.

Note: As described in the Study Population section in the synopsis, before entering the trial, the medical team will present other available experimental therapies to the patient for her consideration.

SUBJECT EXCLUSION CRITERIA

1. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the non-myeloablative, lymphodepleting induction regimen on the fetus or infant. (Note: Pregnancies occurring in patients with Ovarian cancer are very rare, but possible. For this reason, ELIM has decided to retain the sections dealing with possible cases of pregnancy during the study.)
2. Systemic steroid therapy required (patients who require replacement therapy for adrenal insufficiency may be enrolled if steroid treatment dose do not exceed 10 mg of prednisone or equivalent).
3. Active systemic infections, coagulation disorders or other active major medical illnesses of the cardiovascular, respiratory or immune system, as evidenced by a positive stress thallium or comparable test, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
4. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease and AIDS).
5. Opportunistic infections (the experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities.)
6. History of severe immediate hypersensitivity reaction to any of the agents used in this study , including history of an anaphylactic reaction to penicillin or gentamicin
7. History of coronary revascularization or ischemic heart disease.
8. Any patient known to have an LVEF less than or equal to 50 percent.
9. Documented LVEF of less than or equal to 50 percent tested in patients with clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block
10. Documented FEV1 and DLCO (relative to predicted) less than or equal to 60 percent.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Metastatic Malignant Ovarian Cancer
Enrollment: 15 (Estimated)
Dates: Start 2018-01-21 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Objective Tumor responses | 3 years
  Radiological follow up via CT to determine the sum of complete Responders (CR) + Partial Responders (PR) +Stable Disease (SD) as assessment by RECICT 1.1
Assess adverse events using NCI CTCAE V.4.03 during treatment and follow up | 3 years
  adverse events will be assess using MCI CTCAE V.4.03 during treatment and follow up

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years
  Overall survival is defined as the time from study entry until death from any cause
Response Rate( RR) | 3 years
  Radiological follow up via CT to determine the sum of complete responders (CR) + Partial responders (PR) as assessed by RECICT 1.1
Progression Free Survival (PFS) | 3 years
  Progression free survival according to RECICT 1.1
Quality of Life (QoL) | 3 years
  assessment of Quality of Life (QoL) using disease specific modules of the EORTC QLQ-C30 (version 3.0)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Schachter, Prof., Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided
to be considered